CLINICAL TRIAL: NCT05220371
Title: Influence of Specific Collagen Peptides on Parameters of Biomechanical and Systemic Recovery After Exercise-induced Muscle Damage
Brief Title: Influence of Specific Collagen Peptides on Recovery After Exercise Induced Muscle Damage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vienna (Other)
Collaborators: CRI Collagen Research Institute GmbH (Unknown)
Responsible Party: Principal Investigator, Daniel König, Univ.-Prof. Dr. med. Daniel König, University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 00765
Record Dates: First submitted 2022-01-28; First posted 2022-02-02 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Recovery
Keywords: Collagen peptides; Concurrent training; Ultrasound; MVC; RFD
MeSH Terms: interventions — Collagen

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind, randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collagen (Experimental): 15g of collagen peptides ingested daily
  Interventions: Dietary Supplement: Collagen; Other: Concurrent training
- Placebo (Placebo Comparator): 15g of Placebo ingested daily
  Interventions: Other: Concurrent training

INTERVENTIONS:
Dietary Supplement: Collagen — Participants ingest 15 grams of either specific collagen peptides or Placebo daily
  Arms: Collagen
Other: Concurrent training — Both arms undergo a 12-week trainingintervention 3x/week

SUMMARY:
The present study aims at investigating the potential influence of specific collagen peptides on recovery after exercise induced muscle damage with focus on long-term effects.

ELIGIBILITY:
Inclusion Criteria:

* No subjective symptoms during physical exertion
* Stable weight and dietary behaviour
* Body Mass Index (BMI) between 18.5 and 24.9
* No extensive strength/endurance sports so far (less than 3 h/week)
* No complaints during strenuous physical activity

Exclusion Criteria:

* Circumstances that impair/prevent sporting activity (e.g. chronic heart disease, arrhythmia, heart valve disease, arthritis etc.)
* Intolerance/aversion to animal protein
* Arterial hypertension (high blood pressure) (syst > 200 mmHg and/or diast > 105 mmHg) at rest
* Presence of insulin-dependent diabetes mellitus
* Liver and/or kidney disease that precludes a high protein load
* Collagen supplementation or regular intake of other dietary supplements in the last 6 months.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in maximal voluntary contraction (MVC) | Baseline (pre, post, 24 hours, 48 hours) and after 12 weeks (pre, post, 24 hours, 48 hours)
  Measured by isokinetic dynamometer
Change in rate of force development (RFD) | Baseline (pre, post, 24 hours, 48 hours) and after 12 weeks (pre, post, 24 hours, 48 hours)
  Measured by isokinetic dynamometer
Change in countermovement jump height (CMJ) | Baseline (pre, post, 24 hours, 48 hours) and after 12 weeks (pre, post, 24 hours, 48 hours)
  Measured by force plate
Change in subjective pain score | Baseline (pre, post, 24 hours, 48 hours) and after 12 weeks (pre, post, 24 hours, 48 hours)
  Measured by visual analogue scale
Change in Achilles tendon cross-sectional area | Baseline and after 12 weeks
  Measured by ultrasound
Change in Vastus Lateralis fibre length | Baseline (pre, post, 24 hours, 48 hours) and after 12 weeks (pre, post, 24 hours, 48 hours)
  Measured by ultrasound
Change in collagen related blood markers | Baseline (pre, post, 2 hours, 24 hours, 48 hours) and after 12 weeks (pre, post, 2 hours, 24 hours, 48 hours)
  Measured by blood analysis
Change in Achilles tendon echo intensity | Baseline and after 12 weeks
  Measured by ultrasound
Change in Vastus Lateralis echo intensity | Baseline and after 12 weeks
  Measured by ultrasound
Change in body composition parameters (fat mass, fat-free mass, extracellular mass, body cell mass) | Baseline and after 12 weeks
  Measured by bioelectrical impedance analysis

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Koenig, Prof. Dr., Principal Investigator — University of Vienna, Institute of Sport Science
Locations (1):
- University of Vienna, Institute of Sport Science, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bischof K, Stafilidis S, Bundschuh L, Oesser S, Baca A, Konig D. Reduction in systemic muscle stress markers after exercise-induced muscle damage following concurrent training and supplementation with specific collagen peptides - a randomized controlled trial. Front Nutr. 2024 Mar 25;11:1384112. doi: 10.3389/fnut.2024.1384112. eCollection 2024. PMID 38590831
- [Derived] Bischof K, Stafilidis S, Bundschuh L, Oesser S, Baca A, Konig D. Influence of specific collagen peptides and 12-week concurrent training on recovery-related biomechanical characteristics following exercise-induced muscle damage-A randomized controlled trial. Front Nutr. 2023 Nov 16;10:1266056. doi: 10.3389/fnut.2023.1266056. eCollection 2023. PMID 38035363